CLINICAL TRIAL: NCT02270281
Title: Dexmedetomidine Improve Microcirculatory Alterations in Initial Resuscitated Septic Shock Patients
Brief Title: Dexmedetomidine on Microcirculation in Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, MD, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014ZDSYLL093.0
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Septic Shock
Keywords: Sepsis; Sedation; Microcirculation; Dexmedetomidine
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexmedetomidine (Other): Before dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine 0.7 Mcg/kg/h

INTERVENTIONS:
Drug: Dexmedetomidine 0.7 Mcg/kg/h — CIF 0.7mcg/kg/h
  Other Names: Dexmedetomidine

SUMMARY:
Dexmedetomidine was found might be beneficial to sepsis. Dexmedetomidine were found to improve microcirculation in sepsis animal studies and non-sepsis patients. However, the effect of dexmedetomidine on microcirculation in septic shock patients is unknown.

DETAILED DESCRIPTION:
Septic shock is characterized by significant decline in vascular response and relative hypovolemia. Fluids and exogenous catecholamines are mainstay. However, even after initial resuscitation, microcirculatory dysfunctions still exist, and represent a direct physiologic link to organ failure and death. Therefore, therapeutic strategies aiming at improving microcirculation are performed.

Dexmedetomidine was found might be beneficial to sepsis. Dexmedetomidine were found to improve microcirculation in sepsis animal studies and non-sepsis patients. However, the effect of dexmedetomidine on microcirculation in septic shock patients is unknown.

Based on the hypothesis that dexmedetomidine might improve microcirculation in initial resuscitated septic shock patients, the study was to investigate the effects of dexmedetomidine on microcirculation in early septic shock patients despite initial resuscitation. Meanwhile, to observe the possible mechanism of the effect, the correlation between dexmedetomidine dose and microcirculatory parameters as well as catecholamine level were performed.

ELIGIBILITY:
Adult patients who met the following inclusion criteria were enrolled in the study: 1) With septic shock defined by the 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference for less than 24 hours.

2) After initial fluid resuscitation but still requiring norepinephrine to maintain arterial pressure or hyperlactacidemia.

3) Need ongoing analgesia and sedation. 4) Using advanced invasive hemodynamic monitoring techniques.

Exclusion criteria were as follows:

1. age less than 18 years.
2. pregnancy.
3. heart rate less than 55 beats per minute.
4. acute hepatic failure
5. brain injury.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Perfused vascular density | One hour
  Perfused vascular density was calculated by multiplying vessel density by the proportion of perfused vessels

SECONDARY OUTCOMES:
Microcirculatory flow index | One hour
  Based on the major type of flow in all quadrants were determined with a semi-quantitative methodology
Total vascular density | One hour
  Vascular density was calculated by the number of vessels crossing these lines

CONTACTS AND LOCATIONS:
Overall Officials: fengmei Guo, MD,PhD, Study Director — Southeast University
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Result] Massey MJ, Hou PC, Filbin M, Wang H, Ngo L, Huang DT, Aird WC, Novack V, Trzeciak S, Yealy DM, Kellum JA, Angus DC, Shapiro NI; ProCESS investigators. Microcirculatory perfusion disturbances in septic shock: results from the ProCESS trial. Crit Care. 2018 Nov 20;22(1):308. doi: 10.1186/s13054-018-2240-5. PMID 30458880
- [Result] Hernandez G, Tapia P, Alegria L, Soto D, Luengo C, Gomez J, Jarufe N, Achurra P, Rebolledo R, Bruhn A, Castro R, Kattan E, Ospina-Tascon G, Bakker J. Effects of dexmedetomidine and esmolol on systemic hemodynamics and exogenous lactate clearance in early experimental septic shock. Crit Care. 2016 Aug 2;20(1):234. doi: 10.1186/s13054-016-1419-x. PMID 27480413
- [Result] Geloen A, Chapelier K, Cividjian A, Dantony E, Rabilloud M, May CN, Quintin L. Clonidine and dexmedetomidine increase the pressor response to norepinephrine in experimental sepsis: a pilot study. Crit Care Med. 2013 Dec;41(12):e431-8. doi: 10.1097/CCM.0b013e3182986248. PMID 23963131
- [Result] Morelli A, Sanfilippo F, Arnemann P, Hessler M, Kampmeier TG, D'Egidio A, Orecchioni A, Santonocito C, Frati G, Greco E, Westphal M, Rehberg SW, Ertmer C. The Effect of Propofol and Dexmedetomidine Sedation on Norepinephrine Requirements in Septic Shock Patients: A Crossover Trial. Crit Care Med. 2019 Feb;47(2):e89-e95. doi: 10.1097/CCM.0000000000003520. PMID 30394918
- [Result] Miranda ML, Balarini MM, Bouskela E. Dexmedetomidine attenuates the microcirculatory derangements evoked by experimental sepsis. Anesthesiology. 2015 Mar;122(3):619-30. doi: 10.1097/ALN.0000000000000491. PMID 25313879
- [Result] Yeh YC, Wu CY, Cheng YJ, Liu CM, Hsiao JK, Chan WS, Wu ZG, Yu LC, Sun WZ. Effects of Dexmedetomidine on Intestinal Microcirculation and Intestinal Epithelial Barrier in Endotoxemic Rats. Anesthesiology. 2016 Aug;125(2):355-67. doi: 10.1097/ALN.0000000000001135. PMID 27111533
- [Derived] Xu J, Wang Y, Shu C, Chang W, Guo F. Dexmedetomidine Improves Microcirculatory Alterations in Patients With Initial Resuscitated Septic Shock. J Intensive Care Med. 2025 Feb;40(2):137-144. doi: 10.1177/08850666241267860. Epub 2024 Aug 28. PMID 39193773